CLINICAL TRIAL: NCT02568852
Title: Comparison of Coagulation Factors During Laparoscopic Cholecystectomy With General Anesthesia and Spinal-epidural Anesthesia:Prospective Randomized Trials
Brief Title: Comparison of Coagulation Factors During Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lütfiye Nuri Burat Government Hospital (Other Government)
Responsible Party: Principal Investigator, TURGUT DONMEZ, General Surgeon, MD, Lütfiye Nuri Burat Government Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: lutfiyeETD
Record Dates: First submitted 2015-10-01; First posted 2015-10-06 (Estimated); Results first posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-05

CONDITIONS: Gall Stone Disease; Polyp
Keywords: D-dimer; Fibrinogen; Laparoscopic cholecystectomy
MeSH Terms: conditions — Polyps | interventions — Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group 1 (Active Comparator): Laparoscopic cholecystectomy in general anaesthesia
  Interventions: Procedure: Combined anaesthesia
- group 2 (Active Comparator): Laparoscopic cholecystectomy in combined anaesthesia (Spino epidural).
  Interventions: Procedure: General anaesthesia

INTERVENTIONS:
Procedure: Combined anaesthesia — Laparoscopic cholecystectomy under 10 mmHg pressure
  Arms: group 1
Procedure: General anaesthesia — Laparoscopic cholecystectomy under 10 mmHg pressure
  Arms: group 2

SUMMARY:
Pneumoperitoneum is formed with CO2 during laparoscopic abdominal operations. Effect of pneumoperitoneum on coagulation factors is not well known. In our study the investigators aimed to compare the general anesthesia(GA) and combined spinal-epidural anesthesia (CA) during laparoscopic cholecystectomy(LC) with effect on coagulation factors.

Fifty patients will be randomly assigned to either the Laparoscopic cholecystectomy under Combined anaesthesia (25 patients) or Laparoscopic cholecystectomy under general anaesthesia (25 patients). All patients has symptomatic gall stone disease or polyp of gall bladder.

DETAILED DESCRIPTION:
Objective of study : The aim of this study was to compare general anesthesia (GA) and combined (epidural and spinal) anesthesia (CA) for laparoscopic cholecystectomy(LC).Laparoscopic cholecystectomies are usually performed under general anesthesia. Studies involving cholecystectomies with regional anesthesia recently published. During regional anesthesia pneumoperitoneum is performed with lower pressure(10mmHg CO2). Patients can not tolerate higher intraabdominally pressure. Thera are very few studies involving the effect of pneumoperitoneum on coagulation factors. In our study the investigators separate the patients into 2 groups. Group1:10 mmHg pressure, laparoscopic cholecystectomy under general anesthesia ; Group2 : 10 mmHg pressure, laparoscopic cholecystectomy under Combined Spinal-Epidural Anesthesia The investigators performed standard conventional laparoscopic cholecystectomy procedure with 10mmHg pressure in both groups. The investigators aimed to investigate Prothrombin Time(PT), activated partial thromboplastin time(aPTT), thrombin time(TT), D-dimer and fibrinogen levels preoperative, postoperative 1st hour and 24th hour respectively.

ELIGIBILITY:
Inclusion Criteria:

* Gall bladder stone
* Gall bladder polyp

Exclusion Criteria:

* Pregnancy
* Malignancy
* Children
* Acute cholecystitis
* Vertebral deformities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Donmez, Surgeon, Principal Investigator — Lutfiye Nuri Burat Goverment Hospital
Locations (1):
- Lutfiye NBGH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
yes

REFERENCES:
- [Background] Ntourakis D, Sergentanis TN, Georgiopoulos I, Papadopoulou E, Liasis L, Kritikos E, Tzardis P, Laopodis V. Subclinical activation of coagulation and fibrinolysis in laparoscopic cholecystectomy: do risk factors exist? Int J Surg. 2011;9(5):374-7. doi: 10.1016/j.ijsu.2011.02.011. Epub 2011 Mar 1. PMID 21371576
- [Background] Frantzides CT, Welle SN, Ruff TM, Frantzides AT. Routine anticoagulation for venous thromboembolism prevention following laparoscopic gastric bypass. JSLS. 2012 Jan-Mar;16(1):33-7. doi: 10.4293/108680812X13291597716906. PMID 22906327

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Laparoscopic cholecystectomy under general anaesthesia
- Group 2: Laparoscopic cholecystectomy under combined anaesthesia (Spino epidural).
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Laparoscopic cholecystectomy in under 10 mmHg pneumoperitoneum
- Group 2: Laparoscopic cholecystectomy in under 14 mmHg pneumoperitoneum
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Full Range); unit: years] | 46 [19 to 69] | 52 [27 to 79] | 48 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  Turkey | 25 | 25 | 50
ASA(American Society of Anesthesiologists ) scores [Median (Full Range); unit: Scores on a scale(min:1 and max:6)] — ASA scores:ASA 1(better) and ASA VI(worse) ASA I:A normal healthy patient ASA II:A patient with mild systemic disease ASA III:A patient with severe systemic disease ASA IV:A patient with severe systemic disease that is a constant threat to life ASA V:A moribund patient who is not expected to survive without the operation ASA VI:A declared brain-dead patient whose organs are being removed for donor purposes
  Scores on a scale(min:1 and max:6) | 1 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
BMI [Median (Standard Deviation); unit: kg/m^2] — BMI:Body Mass Index
  kg/m^2 | 28.1 (4.0) | 28.2 (3.5) | 28.15 (3.72)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Operation
Description: group1 and group 2(Duration of Operation)
Time Frame: up to 2 hours
Population: All patients have gall bladder disease who are between 18-80 years old.
Measure: Mean (Full Range); unit: minutes
Groups:
- Group 1: Laparoscopic cholecystectomy in general anaesthesia
  Combined anaesthesia: 10 mmHg pressure, laparoscopic cholecystectomy under combined spinal epidural anaesthesia
- Group 2: Laparoscopic cholecystectomy in combined anaesthesia (Spino epidural).
  General anaesthesia: 10 mmHg pressure, laparoscopic cholecystectomy under general anesthesia
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
minutes | 54 [45 to 80] | 65 [53 to 92]

2. Secondary Outcome: Fibrinogen Level
Description: A soluble plasma glycoprotein, that is converted by thrombin into fibrin during blood clot formation
Time Frame: pre-operative
Population: All patients have gall bladder disease who are between 18-80 years old.
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
mg/dL | 219 [138 to 318] | 261 [87 to 395]

3. Secondary Outcome: Fibrinogen Level
Description: A soluble plasma glycoprotein, that is converted by thrombin into fibrin during blood clot formation
Time Frame: Post-operative 1 st hour
Population: All patients have gall bladder disease who are between 18-80 years old.
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
mg/dL | 253 [214 to 382] | 320 [171 to 495]

4. Secondary Outcome: Fibrinogen Level
Description: A soluble plasma glycoprotein, that is converted by thrombin into fibrin during blood clot formation
Time Frame: Post-operative 24th hour
Population: All patients have gall bladder disease who are between 18-80 years old.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
mg/dL | 352 [258 to 496] | 421 [250 to 760]

5. Secondary Outcome: PT(Prothrombin Time)
Description: measures of the extrinsic pathway of coagulation
Time Frame: pre-operative
Population: All patients have gall bladder disease who are between 18-80 years old.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
seconds | 11.94 (0.64) | 11.78 (0.75)

6. Secondary Outcome: PT(Prothrombin Time)
Description: measures of the extrinsic pathway of coagulation
Time Frame: Post-operative 1st hour
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
seconds | 12.1 (0.53) | 12.69 (0.84)

7. Secondary Outcome: PT(Prothrombin Time)
Description: measures of the extrinsic pathway of coagulation
Time Frame: Post-operative 24th hours
Population: All patients have gall bladder disease who are between 18-80 years old.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
seconds | 12.43 (0.86) | 13.63 (1.07)

8. Secondary Outcome: D-Dimer
Description: A fibrin degradation product (or FDP) present in the blood after a blood clot is degraded by fibrinolysis
Time Frame: pre-operative
Population: All patients have gall bladder disease who are between 18-80 years old.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
mg/L | 0.31 (0.08) | 0.34 (0.10)

9. Secondary Outcome: D-Dimer
Description: A fibrin degradation product (or FDP) present in the blood after a blood clot is degraded by fibrinolysis
Time Frame: Post-operative 1st hour
Population: All patients have gall bladder disease who are between 18-80 years old.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
mg/L | 0.56 (0.22) | 1.06 (0.7)

10. Secondary Outcome: D-Dimer
Description: A fibrin degradation product (or FDP) present in the blood after a blood clot is degraded by fibrinolysis
Time Frame: Post-operative 24th hours
Population: All patients have gall bladder disease who are between 18-80 years old.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
mg/L | 0.91 (0.34) | 1.61 (0.95)

11. Secondary Outcome: aPTT(Activated Partial Thromboplastin Time)
Description: measures of the intrinsic pathway of coagulation
Time Frame: pre-operative
Population: All patients have gall bladder disease who are between 18-80 years old.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
seconds | 22.80 (1.48) | 25.0 (2.86)

12. Secondary Outcome: aPTT(Activated Partial Thromboplastin Time)
Description: measures of the intrinsic pathway of coagulation
Time Frame: Post-operative 1st hour
Population: All patients have gall bladder disease who are between 18-80 years old.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
seconds | 23.42 (1.54) | 25.25 (2.35)

13. Secondary Outcome: aPTT(Activated Partial Thromboplastin Time)
Description: measures of the intrinsic pathway of coagulation
Time Frame: Post-operative 24th hours
Population: All patients have gall bladder disease who are between 18-80 years old.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
seconds | 24.54 (2.16) | 26.92 (2.92)

14. Secondary Outcome: Thrombin Time(TT)
Description: measures of the extrinsic and intrinsic pathway of coagulation
Time Frame: pre-operative
Population: All patients have gall bladder disease who are between 18-80 years old.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
seconds | 19.88 (1.58) | 20.57 (2.12)

15. Secondary Outcome: Thrombin Time(TT)
Description: measures of the extrinsic and intrinsic pathway of coagulation
Time Frame: Post-operative 1st hour
Population: All patients have gall bladder disease who are between 18-80 years old.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
seconds | 17.78 (0.74) | 17.61 (1.02)

16. Secondary Outcome: Thrombin Time(TT)
Description: measures of the extrinsic and intrinsic pathway of coagulation
Time Frame: Post-operative 24th hours
Population: All patients have gall bladder disease who are between 18-80 years old.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 25
seconds | 16.06 (1.05) | 16.01 (0.72)

ADVERSE EVENTS:
Time Frame: up to 24 weeks
Description: In this time period, hypotension,urinary retention,nausea and headache were observed.
Groups:
- Group 1: Laparoscopic cholecystectomy in under general anaesthesia.(10 mmHg CO2 pneumoperitoneum)
- Group 2: Laparoscopic cholecystectomy in under spinal epidural anaesthesia.(10 mmHg CO2 pneumoperitoneum)
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 5/25 | 5/25
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=25) | Group 2 (N=25)
Hypotension (Cardiac disorders) | 1 (1) | 2 (2)
urinary retension (Renal and urinary disorders) | 0 (0) | 1 (1)
Nausea/vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No